CLINICAL TRIAL: NCT00888979
Title: Pilot Study of Nicotine Replacement for Smoking Cessation During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: UConn Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONCK002885HU; H09-183-2 (Other: Hartford Hospital)
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking Cessation during Pregnancy; Nicotrol Inhaler
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nicotrol with Behavioral Counseling (Experimental): Nicotrol Inhaler: 10 mg of nicotine per one inhaler cartridge. Inhaler use will substitute the usual smoking pattern
  Interventions: Drug: Nicotrol Inhaler

INTERVENTIONS:
Drug: Nicotrol Inhaler — 10 mg of nicotine per one inhaler cartridge. Inhaler use will substitute the usual smoking pattern

SUMMARY:
We plan to examine the feasibility, acceptability, preliminary quit rates, overall nicotine exposure and adverse effects of the nicotine inhaler for smoking cessation in pregnancy.

DETAILED DESCRIPTION:
Subjects in this pilot study are healthy pregnant women who wish to quit smoking. They will set a quit date and use the nicotine inhaler for 4 weeks. They will receive behavioral counseling in addition to the inhaler for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 13-26 weeks pregnant
* Smoking at least 5 cigarettes per day the preceding 7 days
* Motivated to quit smoking (at least 7 on a 10 pt. scale)
* Able to speak English
* Intend to carry pregnancy to term
* Stable residence

Exclusion Criteria:

* Current drug or alcohol abuse or dependence (other than methadone maintenance
* Twins or multiple gestation
* Unstable psychiatric disorder
* Unstable medical problems
* Known congenital abnormality
* High risk pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2011-05 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Oncken, MD MPH, Principal Investigator — UConn Health
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotrol Inhaler With Behavioral Counseling: Nicotrol Inhaler: 10 mg of nicotine per one inhaler cartridge. Inhaler use will substitute the usual smoking pattern
Period: Overall Study
Arm/Group | Nicotrol Inhaler With Behavioral Counseling
Started | 10
Received the Inhaler/Counseling | 8
Completed | 6
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Nicotrol Inhaler With Behavioral Counseling
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 26 [19 to 38]
Gender [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Days of Inhaler Use
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nicotrol Inhaler With Behavioral Counseling
Number analyzed (Participants) | 6
days | 26.4 (3)

2. Secondary Outcome: Cartridge Use
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: cartridges per day
Arm/Group | Nicotrol Inhaler With Behavioral Counseling
Number analyzed (Participants) | 6
cartridges per day | 2 (1.5)

3. Secondary Outcome: Change in Number of Cigarettes Used Per Day From Baseline to 4 Weeks.
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: reduction in number of CPD
Arm/Group | Nicotrol Inhaler With Behavioral Counseling
Number analyzed (Participants) | 6
reduction in number of CPD | -5.7 (2.3)

ADVERSE EVENTS:
Time Frame: Baseline to delivery, up to 27 weeks)
Arm/Group | Nicotrol Inhaler With Behavioral Counseling
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotrol Inhaler With Behavioral Counseling (N=8)
preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotrol Inhaler With Behavioral Counseling (N=8)
Nausea (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (3)
Lightheadedness (General disorders) | 1 (1)
heartburn (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No